CLINICAL TRIAL: NCT02599012
Title: The Efficacy of Intravenous Iron for the Treatment of Anemia in Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jun Ho Jang, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01-011-001
Record Dates: First submitted 2015-10-07; First posted 2015-11-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Cancer; Anemia
MeSH Terms: conditions — Neoplasms; Anemia | interventions — ferric carboxymaltose

ARMS (1):
- Subjects (Experimental)
  Interventions: Drug: Ferinject®

INTERVENTIONS:
Drug: Ferinject® — intravenous Ferinject 1000mg injection

SUMMARY:
* Multifactorial pathogenesis is involved in anemia of cancer patients and defining the causes of anemia is not always simple.
* Currently, treatment options available for anemia in cancer patients include red blood cell (RBC) transfusion, erythropoietin stimulating agent (ESA), and iron supplementation, accompanying considerable pros and cons for each treatment.
* Previous studies have demonstrated benefit when treating with IV iron in combination with ESA and, more recently, evidence is emerging to suggest a role for IV iron alone.
* In this study, investigator will assess the efficacy of intravenous iron for the treatment of anemia in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who diagnosed with solid cancer or lymphoma
* Subjects who are under anti-cancer therapy at enrollment or has finished anti-cancer therapy within 2 months before enrollment

  * anticancer therapy: "chemotherapy", and/or "chemotherapy + radiotherapy", and/or "target agent"
* Subjects whose Hb level is 8.0-10.5g/dL, or who experienced a drop of Hb by 2g/dL or more during anti-cancer treatment

Exclusion Criteria:

* Subjects who received iron (oral or iv), ESA, dialysis within 4 weeks before enrollment
* Subjects with uncontrolled infection
* Subjects with ongoing bleeding
* Deteriorated organ function
* poor performance state (ECOG 3-4)
* Subjects whose disease involves bone marrow
* Ferritin > 800 ng/ml and Transferrin saturation(TSAT) ≥ 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09-12 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Hemoglobin response | visit 4th after Ferinject injection

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Irwon-ro ,Kangnam-gu, South Korea

REFERENCES:
- [Derived] Jang JH, Kim Y, Park S, Kim K, Kim SJ, Kim WS, Jung CW, Lee J, Lee SH. Efficacy of intravenous iron treatment for chemotherapy-induced anemia: A prospective Phase II pilot clinical trial in South Korea. PLoS Med. 2020 Jun 8;17(6):e1003091. doi: 10.1371/journal.pmed.1003091. eCollection 2020 Jun. PMID 32511251
- See also: Iron deficient erythropoiesis might play key role in development of anemia in cancer patients. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Iron+deficient+erythropoiesis+might+play+key+role+in+development+of+anemia+in+cancer+patients